CLINICAL TRIAL: NCT07344441
Title: Accuracy of Patient Specific 3D Printed Titanium Plates Versus 3D Milled Titanium Plates in Genioplasty Orthognathic Surgeries. A Randomized Controlled Clinical Trial
Brief Title: Accuracy of Patient Specific 3D Printed Titanium Plates Versus Milled Titanium Plates in Genioplasty Orthognathic Surgeries.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina ElHadidi Sobhi Ramzi Michael, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: patient specific genioplasty
Record Dates: First submitted 2025-12-26; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Accuracy of 3D Printed Titanium Plates Versus 3D Milled Titanium Plates in Genioplasty Orthognathic Surgery; Patient Specific Genioplasty; Accuracy of 3D Printed Titanium Plates Versus 3D Milled Titanium Plates in Genioplasty
Keywords: accuracy of 3D printed titanium plates versus 3D milled titanium plates in genioplasty; patient specific genioplasty; patient specific 3D printed titanium plates genioplasty; patient specific 3D milled titanium plates genioplasty; genioplasty orthognathic surgery
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: the treatment include fixing the chin in genioplasty orthognathic surgery with 3D printed patient specific titanium plates
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Experimental : genioplasty using 3D printed patient specific titanium plates (study group) The first treatment plan includes fixing the chin with 3D printed patient specific titanium plates in genioplasty orthognathic surgery
  Interventions: Procedure: genioplasty using 3D printed patient specific titanium plates (study group)
- control Group (Experimental): Experimental : genioplasty using 3D milled patient specific titanium plates (study group) The second treatment plan includes fixing the chin with 3D milled patient specific titanium plates in genioplasty orthognathic surgery
  Interventions: Procedure: genioplasty using 3D milled patient specific titanium plates (control group)

INTERVENTIONS:
Procedure: genioplasty using 3D printed patient specific titanium plates (study group) — genioplasty using 3D printed patient specific titanium plates (study group) the treatment plan includes fixing the chin with 3D printed patient specific titanium plates in genioplasty orthognathic surgery
  Arms: Study Group
Procedure: genioplasty using 3D milled patient specific titanium plates (control group) — genioplasty using 3D milled patient specific titanium plates (control group) The treatment plan includes fixing the chin with 3D milled patient specific titanium plates in genioplasty orthognathic surgery
  Arms: control Group

SUMMARY:
To assess accuracy of patient specific 3D printed titanium plates versus 3D milled titanium plates in genioplasty orthognathic surgery

DETAILED DESCRIPTION:
the first treatment include treating patients with 3D printed titanium plates while the second treatment include treating patients with 3D milled titanium plates in genioplasty orthognathic surgery and assess the accuracy between the two treatments

ELIGIBILITY:
Inclusion Criteria:

1. Patients with dentofacial disharmony and misalignment requiring bimaxillary orthognathic surgeries.
2. Patients with no signs or symptoms of active TMDs.
3. Highly motivated patients.

Exclusion Criteria:

1. Patients who refused to be included in the research.
2. Patients with systemic diseases that may hinder the normal healing process or render the patient not fitting for general anaesthesia.
3. Patients with intra-bony lesions or infections that may retard the osteotomy healing.
4. Patients with systemic condition contraindicating with the surgical procedure as uncontrolled diabetes

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-11-01 (Estimated); Primary Completion 2027-05-10 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of manufacturing of the patient specific 3D printed titanium plates versus milled titanium plates in genioplasty | immediately postoperative
  Accuracy of manufacturing of the patient specific customized 3D printed titanium plates in the study group versus milled titanium plates in the control group in genioplasty measure The skull base in the virtual surgical plan was superimposed using point-based matching ICP registration using anatomical reference points, followed by manual surface-based registration to surface best fit with the skull base in the actual post-operative CBCT scans.
  the measurement tool is CBCT scans superimposition in mm

SECONDARY OUTCOMES:
stability of manufacturing of the patient specific 3D printed titanium plates versus milled titanium plates in genioplasty | 6 months postoperative
  stability of manufacturing of the patient specific customized 3D printed titanium plates in the study group versus milled titanium plates in the control group in genioplasty The skull base in the virtual surgical plan was superimposed using point-based matching ICP registration using anatomical reference points, followed by manual surface-based registration to surface best fit with the skull base in the actual 6 months post-operative CBCT scans.
  the measurement tool is CBCT scans superimposition in mm

OTHER OUTCOMES:
Soft tissue dehiscence | 2 months postoperatively
  measurement of the amount of dehiscence and exposure of the plate and bone vertically and horizontally by periodontal probe the measurement tool is periodontal probe
Patient satisfaction | at the recruitment visit and 6 months postoperative
  by Condition specific questionnaire asking the patient with score for satisfaction of the result and to assess the quality of life A self-administered OQLQ translated into Arabic will be used to assess quality of life at the recruitment visit and six months after the surgery. Questions 1, 7, 10, 11, and 14 will be about facial aesthetics and appearance, questions 2 to 6 will be about oral function, questions 8, 9, 12, and 13 will be about the awareness of the deformity, and questions 15 to 22 will about the social aspect of the deformity.
  The questionnaire contains 22 questions, and each question has score from 1 to 4, so each patient will have a score from 22 to 88.
  the measument tool is questionaire chart

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mounir Shaker, Study Chair — Cairo University; Rofaida Atef Abaas, Study Director — Cairo University; Mohamed Ali Zain El Abdeen Abd El Wahab, Study Director — Cairo University

REFERENCES:
- [Background] Hanafy M, Akoush Y, Abou-ElFetouh A, Mounir RM. Precision of orthognathic digital plan transfer using patient-specific cutting guides and osteosynthesis versus mixed analogue-digitally planned surgery: a randomized controlled clinical trial. Int J Oral Maxillofac Surg. 2020 Jan;49(1):62-68. doi: 10.1016/j.ijom.2019.06.023. Epub 2019 Jun 29. PMID 31262680
- [Background] Levine JP, Patel A, Saadeh PB, Hirsch DL. Computer-aided design and manufacturing in craniomaxillofacial surgery: the new state of the art. J Craniofac Surg. 2012 Jan;23(1):288-93. doi: 10.1097/SCS.0b013e318241ba92. PMID 22337427
- [Background] Kusnoto B. Two-dimensional cephalometry and computerized orthognathic surgical treatment planning. Clin Plast Surg. 2007 Jul;34(3):417-26. doi: 10.1016/j.cps.2007.04.005. PMID 17692701
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17692701/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22337427/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31262680/